CLINICAL TRIAL: NCT05957913
Title: Effects of Antiviral Therapies on Epstein-Barr Virus Replication
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Solving MS (Unknown)
Responsible Party: Principal Investigator, Michael, Levy M.D.,Ph.D., Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023P000828
Record Dates: First submitted 2023-06-28; First posted 2023-07-24 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir; Emtricitabine

STUDY DESIGN:
Intervention Model Description: The study design will be an open-label single arm study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): After a one-month baseline period where patients will not take any study drug, all patients will receive Truvada (tenofovir/emtricitabine) for three months. The study drug will be Truvada (tenofovir/emtricitabine), an antiviral drug that is approved by the Food & Drug Administration (FDA) for the treatment of chronic hepatitis B virus and for the treatment and prevention of human immunodeficiency virus (HIV) infection. The study drug will be administered at the standard dose used for the treatment and prevention of HIV (300mg tenofovir disoproxil fumarate, 200mg emtricitabine). Since extensive safety and tolerability data already exists for this standard dose, the selection of this dose also allows us to use existing data to inform strategies for safety and tolerability monitoring to minimize risk, as detailed in the study design.
  Interventions: Drug: Truvada (tenofovir/emtricitabine)

INTERVENTIONS:
Drug: Truvada (tenofovir/emtricitabine) — Doses and route of administration of the study drug will be kept the same as for the FDA-approved indication of HIV-1 prevention in healthy individuals. The study drug is not FDA-approved for the treatment of multiple sclerosis.
  Other Names: TDF

SUMMARY:
This research study is being performed to find out if Truvada (tenofovir/emtricitabine), an antiviral drug with activity against the Epstein Barr virus (EBV), can reduce EBV levels in saliva and blood in people with multiple sclerosis (MS). A second goal is to find out if Truvada (tenofovir/ emtricitabine) is safe and tolerable in people with MS.

DETAILED DESCRIPTION:
The proposed trial is built on the premise that multiple sclerosis (MS) is, in part, triggered by infection with the human herpesvirus Epstein Barr virus (EBV), and that targeting the virus could be a more effective and safer strategy for MS treatment than immunomodulation or immunosuppression alone. The evidence supporting a causal role for EBV in MS initially came from epidemiological studies that showed similarities in the distribution of infectious mononucleosis and MS, a 2-3 fold increased MS risk among individuals with a clinical history of infectious mononucleosis, and by compelling evidence that MS rarely, if ever, develops in individuals who are not infected with EBV. Furthermore, in a longitudinal study based on the Department of Defense Serum Repository with samples from over 7 million young adults free of MS, individuals who were EBV-seronegative at baseline did not develop symptoms of MS until at least several months after EBV seroconversion, and high serum antibody titers against the EBV-encoded nuclear antigen-1 were associated with an over 30-fold increase in MS risk.

Antiviral agents repurposed from treating other herpesviruses, like acyclovir or valacyclovir, have had minimal clinical efficacy against EBV in studies for infectious mononucleosis and multiple sclerosis. Prodrugs of tenofovir, such as tenofovir disoproxil fumarate (TDF), are significantly more potent inhibitors of EBV replication in cell culture than other drugs that have been clinically ineffective for EBV. TDF is a safe drug used clinically for HIV pre-exposure prophylaxis (PrEP) in HIV-negative patients as the drug Truvada. Truvada has been widely used since its approval in 2004 for the treatment of human immunodeficiency virus (HIV), and has a well-known safety profile that makes it a good candidates for clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness and ability to comply with all study procedures and availability for the duration of the study
* Age: 18+
* Established diagnosis of multiple sclerosis
* Evidence of Epstein Barr virus (EBV) infection by serological testing for EBV antibodies antibodies (subjects will have EBV testing performed at the pre-screening visit and if serologies are negative, the subjects will be removed from the study)

Exclusion Criteria:

* Pregnancy or lactation
* Known allergic reactions to components of Truvada
* Previous treatment with Truvada or Descovy
* Unknown HIV status (subjects must have completed HIV antigen/antibody and viral load testing within the prior 6 months to being enrolled or have the testing completed at the pre-screening visit)
* Active or latent hepatitis B (HBV) (subjects must have completed HBV serologies - HbsAg, anti-HBs, and anti-HBc - within the prior 6 months to being enrolled or have the testing completed at the pre-screening visit)
* Current symptoms of severe, progressive, or uncontrolled renal, hematologic, gastrointestinal, pulmonary, cardiac, or neurologic disease, or other medical conditions that, in the opinion of the investigator, might place the subject at unacceptable risk for participation in this study
* Creatinine clearance (CrCl) <75mL/min, as calculated by the Cockcroft-Gault equation
* Urine dipstick for protein and glucose, excluding values of "1 +" or greater
* Any history of bone fractures not explained by trauma
* Confirmed Grade 2 or greater hypophosphatemia
* Any Grade 2 or greater toxicity on screening tests and assessments
* Taking a medication with known interactions with Truvada including but not limited to: Acyclovir, valacyclovir, adefovir, cabozantinib, carbamazepine, cidofovir, cladribine, cobicistat, diclofenac, multiple non-steroidal antiinflammatories (NSAIDs) or chronic high dose NSAIDs, fosphenytoin or phenytoin, ganciclovir, valganciclovir, oxcarbazepine, phenobarbital, primidone, rifabutin, rifampin, rifapentine, sofosbuvir, tipranavir, or other drugs that significantly affect renal function
* Current treatment with drugs known to affect EBV replication as listed below: Acyclovir, valacyclovir, ganciclovir, valganciclovir, famciclovir, teriflunomide, interferon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2026-06-04 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Epstein Barr virus (EBV) viral load | Change from baseline at three months
  EBV viral load will be quantified in saliva and peripheral blood using a sensitive assay.

SECONDARY OUTCOMES:
Tolerability of Truvada (tenofovir/emtricitabine) | Change from baseline at three months
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]
Fatigue | Change from baseline at three months
  Fatigue will be measured using a standardized survey scale where higher scores indicate more fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Michael Levy, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No